CLINICAL TRIAL: NCT04579263
Title: Assessment of Improvement in Glycemic Control, Weight, and Insulin Sensitivity in Obese Patients After Fecal Microbiota Transplantation (FMT) Against the Background of Glucose-lowering Therapy
Brief Title: Assessment of the Health Improvement of Obese Patients After Fecal Microbiota Transplantation (FMT)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal Research and Clinical Center of Physical-Chemical Medicine (Other)
Collaborators: Endocrinology Research Centre, Moscow (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FMT-D1D2
Record Dates: First submitted 2020-09-22; First posted 2020-10-08 (Actual); Last update posted 2020-10-08 (Actual); Status verified 2020-09

CONDITIONS: Obesity; Familial
MeSH Terms: conditions — Obesity | interventions — Fecal Microbiota Transplantation

STUDY DESIGN:
Intervention Model Description: Two obese patients selected according to the inclusion criteria will undergo fecal microbiota transplantation from a healthy donor with a normal body mass index against the background of glucose-lowering therapy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patient with diabetes mellitus type 1 (T1DM) (Experimental): Treatment by transplantation of fecal microbiota
  Interventions: Other: Fecal microbiota
- Patient with diabetes mellitus type 2 (T2DM) (Experimental): Treatment by transplantation of fecal microbiota
  Interventions: Other: Fecal microbiota

INTERVENTIONS:
Other: Fecal microbiota — Transplantation of fecal microbiota of healthy donor with normal body mass index

SUMMARY:
Search for mechanisms of the effect of fecal microbiota transplantation on patients with obesity

DETAILED DESCRIPTION:
1. To select recipients of fecal samples according to eligibility criteria;
2. To perform fecal microbiota transplantation for patients with obesity;
3. To analyze the efficacy of fecal microbiota transplantation for patients with obesity within six months after therapy.

ELIGIBILITY:
Inclusion Criteria:

* age of patients - from 18 to 75 years, both sexes;
* patients with obesity (body mass index ≥40
* patient's informed consent to perform fecal microbiota transplantation

Exclusion Criteria:

* presence of a concomitant chronic infectious disease or malignancy
* patients with a proven allergy to foods not excluded from the donor's diet
* absence of the patient for one or more intermediate stages of the examination.
* informed refusal to continue therapy

Ages: 40 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 2 (Actual)
Dates: Start 2020-02-15 (Actual); Primary Completion 2020-08-15 (Actual); Study Completion 2020-09-22 (Actual)

PRIMARY OUTCOMES:
Change in insulin sensitivity within FMT, 6 months after FMT] | 6 months after FMT
  participants will undergo euglycaemic glucose clamp study

CONTACTS AND LOCATIONS:
Overall Officials: Elena Ilina, MD, Study Director — Federal Research and Clinical Center of Physical-Chemical Medicine; Marina Shestakova, MD, Study Director — Endocrinology Research Centre, Moscow; Elena Zhgun, PhD, Principal Investigator — Federal Research and Clinical Center of Physical-Chemical Medicine; Elena Pokrovskaya, Principal Investigator — Endocrinology Research Centre, Moscow; Igor Sklyanik, Principal Investigator — Endocrinology Research Centre, Moscow
Locations (2):
- Russia (2):
  - Endocrinology Research Centre, Moscow, Moscow
  - Federal Research and Clinical Center of Physical-Chemical Medicine, Moscow (FRCC PCM), Moscow